CLINICAL TRIAL: NCT04402879
Title: A Prospective Randomized Trial of Prone Positioning Versus Usual Care for Patients With Do-not-intubate Goals of Care and Hypoxemic Respiratory Failure During the Coronavirus SARS-CoV-2 (COVID-19) Pandemic
Brief Title: CORONA (COvid pRONe hypoxemiA): Prone Positioning for Hypoxemic COVID-19 Patients With Do-not-intubate Goals
Acronym: CORONA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Collaborators: Alberta Health services (Other)
Responsible Party: Principal Investigator, Ken Kuljit Parhar, MD, Consultant Intensivist & Clinical Assistant Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB20-0518
Record Dates: First submitted 2020-05-22; First posted 2020-05-27 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-05

CONDITIONS: Severe Acute Respiratory Syndrome Coronavirus 2; COVID-19; Acute Respiratory Distress Syndrome; ARDS; Hypoxemic Respiratory Failure
Keywords: Prone positioning; non-intubated
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome; Respiratory Insufficiency | interventions — Prone Position

STUDY DESIGN:
Intervention Model Description: This is a prospective, unblinded, randomized controlled trial at four (4) medical sites in Calgary, Alberta.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prone Positioning (PP) (Experimental): The intervention for this study is PP. Patients at participating sites allocated to the intervention arm of the study will be prompted by ward nurses and respiratory therapists to assume and maintain a prone position for varying durations, four times per day.
  Interventions: Procedure: Prone Positioning (PP)
- Control - usual management (No Intervention): The control group will consist of standard medical care with no instructions or prompts to change positioning to staff or patients.

INTERVENTIONS:
Procedure: Prone Positioning (PP) — The intervention for this study is PP. Patients at participating sites allocated to the intervention arm of the study will be prompted by ward nurses and respiratory therapists to assume and maintain a prone position for varying durations, four times per day until the occurrence of a primary outcome event or hospital discharge.
  The target duration (dose) of PP is > 8 hours per day for up to 60 days, or until oxygen requirements are < 2 L per minute or < 2 L per minute above baseline home oxygen requirements.
  Arms: Prone Positioning (PP)

SUMMARY:
The purpose of this trial is to determine whether Prone Positioning (PP) improves outcomes for non-intubated hospitalized patients with hypoxemic respiratory failure due to COVID-19, who are not candidates for mechanical ventilation in the ICU. The investigators hypothesize that PP will reduce in-hospital mortality or discharge to hospice, compared with usual care for non-intubated patients with do-not-intubate goals of care with hypoxemic respiratory failure due to probable COVID-19.

DETAILED DESCRIPTION:
As part of the management of COVID-19 related severe ARDS, the World Health Organization (WHO) recommends prone positioned mechanical ventilation. At this time, it is unclear whether there is a role for prone positioning (PP) of non-mechanically ventilated patients.

The objective of this trial is to determine whether PP improves outcomes for non-intubated hospitalized patients with hypoxemic respiratory failure due to COVID-19, who are not candidates for mechanical ventilation in the ICU. The investigators hypothesize that PP will reduce in-hospital mortality or discharge to hospice, compared with usual care for non-intubated patients with do-not-intubate goals of care with hypoxemic respiratory failure due to probable COVID-19.

Patients randomized to the intervention arm will continue with prone positioning until study inclusion criteria are no longer met, discharge from hospital, day 60 in hospital, or until death or discharge to hospice. Daily assessments will occur until day 60 or until the patient is discharged from hospital or is deceased. The investigators anticipate recruitment to be completed within 12 months of starting the trial.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with probable COVID-19. Probable is defined as Influenza like illness (ILI) symptoms OR confirmed COVID-19 exposure AND COVID-19 testing performed. ILI is defined as any one of the following symptoms including: fever, new or worsening cough, coryza, new or worsening dyspnea, or sore throat.
* Goals of care are do-not-intubate (R3 or M1/M2 in Alberta).
* Need for oxygen ≥2 L to maintain SpO2 ≥92%. If the patient is on long-term oxygen, the O2 requirements must be ≥2 L above their baseline.
* Patient can be positioned to and from prone to supine with minimal assistance (maximum one person assistance).

Exclusion Criteria:

* Decreased level of consciousness (Glasgow Coma Scale < 10) or precluding ability to self-reposition.
* Hemodynamic instability (Systolic Blood Pressure < 90 mmHg and or Lactate >5 mmol/L or HR >120, not responsive to fluid resuscitation).
* Complete bowel obstruction.
* Active upper gastrointestinal bleeding.
* Poor neck mobility or patient inability to lie prone comfortably.
* Unstable spine, femur, or pelvic fractures.
* Pregnancy - third trimester.
* Full resuscitation status including ICU and willingness to accept invasive mechanical ventilation (i.e. R1/R2 goals of care).
* Imminent palliation or end of life expected on admission (i.e. C1/C2 goals of care).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 596 (Estimated)
Dates: Start 2020-11-10 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Hospital mortality or discharge to hospice | 60 days
  In-hospital mortality or discharge to hospice at Day 60.

SECONDARY OUTCOMES:
Adverse Events and Serious Adverse Events | 60 days
  An Adverse Event (AE) is any unfavourable or other finding (including clinically significant laboratory tests), symptom or disease occurring during the during of the study, whether or not it is considered to be related to the medicinal (investigational) product, not explicitly classified elsewhere in this protocol, and whether or not it is expected. A Serious Adverse Event (AE) is any unfavourable medical finding (including clinically significant laboratory tests) at any dose that:
  * Results in death (primary outcome)
  * Is life threatening
  * Results in persistent of significant disability or incapacity
  * Requires in in-patient hospitalisation or prolongation of Hospitalisation
Change in SpO2 | 60 days
  Change in SpO2 during each PP session (SpO2 in prone position - SpO2 prior to prone positioning). Clinicians will be asked to record this change for the first proning session per shift (for 12 hour shifts this will result in 2 proning sessions being documented per 24 hour period, and for 8 hour shifts this will result in 3 proning sessions being documented per 24 hour period).
Hospital free days | 60 days
  Number of hospital free days in the 60 days after enrolment.
Admission to ICU | 60 days
  Admission to the Intensive Care Unit.
Intubation and mechanical ventilation | 60 days
  Patient is intubated and requires mechanical ventilation.
Initiation of non-invasive ventilation (NIV) or high-flow nasal oxygen (HFNO). | 60 days
  Patient requires non-invasive ventilation (NIV) or high-flow nasal oxygen (HFNO).
Oxygen-free days | 60 days
  The number of oxygen-free days at Day 60 (censored at discharge).
In-hospital death (time) | 60 days
  Time from admission to all-cause in-hospital death.
Death at 90 days | 90 days
  Death at 90 days.

CONTACTS AND LOCATIONS:
Overall Officials: Ken Parhar, MD, MSc, Principal Investigator — University of Calgary; Jason Weatherald, MD, Principal Investigator — University of Calgary
Locations (4):
- Canada (4):
  - Peter Lougheed Centre (PLC), Calgary, Alberta
  - Foothills Hospital Intensive Care Unit, Calgary, Alberta
  - Rockyview General Hospital, Calgary, Alberta
  - South Health Campus, Calgary, Alberta

REFERENCES:
- [Derived] Weatherald J, Norrie J, Parhar KKS. Awake prone positioning in COVID-19: is tummy time ready for prime time? Lancet Respir Med. 2021 Dec;9(12):1347-1349. doi: 10.1016/S2213-2600(21)00368-4. Epub 2021 Aug 20. No abstract available. PMID 34425072